CLINICAL TRIAL: NCT04229043
Title: Examining the Gastric Emptying Halftime of Water Versus a Carbohydrate in Early Labor
Brief Title: Gastric Emptying of Water and Sports Drink in Labor
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Phillip Hess, Principal Investigator, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2019P001110
Record Dates: First submitted 2020-01-10; First posted 2020-01-14 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Pregnancy; Gastric Emptying
MeSH Terms: interventions — Water

STUDY DESIGN:
Intervention Model Description: Subjects in each group will drink one of two drinks: water or sports drink. We will measure the changing volume in the stomach using ultrasound over the next 60 minutes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Early labor, no analgesia: Sports drink (Active Comparator): Subject will ingest 100 ml of a carbohydrate sports drink
  Interventions: Dietary Supplement: Sports drink
- Early Labor, no analgesia: Water (Placebo Comparator): Subject will ingest 100 ml of water
  Interventions: Dietary Supplement: Water
- Early labor, analgesia: Sports drink (Active Comparator): Subject will ingest 100 ml of a carbohydrate sports drink
  Interventions: Dietary Supplement: Sports drink
- Early labor, analgesia: Water (Placebo Comparator): Subject will ingest 100 ml of water
  Interventions: Dietary Supplement: Water

INTERVENTIONS:
Dietary Supplement: Sports drink — Drink that will be ingested
  Arms: Early labor, analgesia: Sports drink; Early labor, no analgesia: Sports drink
Dietary Supplement: Water — Drink that will be ingested
  Arms: Early Labor, no analgesia: Water; Early labor, analgesia: Water

SUMMARY:
To determine the half time of the emptying of the stomach of women in early labor with and without epidural pain relief when drinking either water or a carbohydrate-based sports drink.

DETAILED DESCRIPTION:
This is a randomized un-blinded study comparing the gastric emptying halftime of water versus a carbohydrate-based sports drink.

Cohorts Women in early labor who have not received pain medication will be enrolled in the study. This will be called the 'unmedicated' group. A second cohort of women who have received an epidural in early labor will be enrolled and studied using identical methods. This will be the 'epidural' group.

Study Intervention Subjects in each group will drink one of two drinks: water or sports drink. The changing volume in the stomach will be measured using ultrasound over the next 60 minutes. Subjects will be asked their degree of hunger on a 10-centimeter visual analogue scale prior to drinking, and for the next two hours at regular intervals. Subjects will be free to consume as per obstetric protocols. The study will be finished once the patient consumes food or drink, feels hunger ≥4/10, or two hours after the sports drink.

Hypothesis The primary hypothesis is that water will empty faster than the sports drink. A second hypothesis is that women with epidural pain relief will have similar gastric halftimes as women without pain medications.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age of 36 weeks or greater
* American Society of Anesthesiology Physical Status 2 or 3
* Induction of labor or early labor (cervical dilation < 6cm)
* Singleton gestation

Exclusion Criteria:

* Recent food ingestion (<3 hours)
* Preeclampsia
* Receiving magnesium sulfate
* Having received narcotics within 12 hours
* Diabetes mellitus
* Multiple gestations
* Active nausea or reflux symptoms

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Subjects must be pregnant, at term, and in early labor
Enrollment: 108 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Gastric emptying half time | 60 minutes
  The time in minutes that half of the volume of the stomach has emptied

SECONDARY OUTCOMES:
Hunger | 60 minutes
  The amount of hunger that the subject feels measured on a visual analogue 10-centimeter line, with the left (0 cm) being labeled 'No Hunger' and the right (10 cm) being labeled 'Maximum hunger'

CONTACTS AND LOCATIONS:
Locations (1):
- Beth Isreal Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No